CLINICAL TRIAL: NCT00201695
Title: Phase II Trial of Pegylated Liposomal Doxorubicin (Doxil), Vincristine, and Dexamethasone (DVd) in Combination With Arsenic Trioxide (Trisenox) in Untreated Patients With Symptomatic Multiple Myeloma
Brief Title: Liposomal Doxorubicin, Vincristine, & Dexamethasone Plus Arsenic Trioxide in Untreated Symptomatic Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0354
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
Keywords: Untreated Patients; Symptomatic
MeSH Terms: conditions — Multiple Myeloma | interventions — liposomal doxorubicin; Vincristine; Dexamethasone; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Doxil® — 40 mg/m2 IV day 1
  Other Names: Doxorubicin HCL liposome injection
Drug: Vincristine — 1.4 mg/m2 (maximum 2 mg) IV day 1
  Other Names: Oncovin
Drug: Dexamethasone — 40 mg PO days 1-4
  Other Names: DVd
Drug: Arsenic Trioxide — 0.25 mg/kg IV over 1-4 hours twice per week, week 1-4 of each cycle (i.e., days 1 and 4; 8 and 11; 15 and 18; 22 and 25)
  Other Names: Trisenox, ATO

SUMMARY:
This study will assess the ability of Doxorubicin, Vincristine and Dexamethasone plus arsenic trioxide to achieve an overall response rate of greater than 60%.

DETAILED DESCRIPTION:
Rationale: The chemotherapy combination of doxorubicin, vincristine and dexamethasone (DVd) has been used with some efficacy in patients with multiple myeloma. However, DVd's efficacy is primarily considered palliative for patients with this condition. The current study adds arsenic trioxide to the DVd combo to assess if all of the treatments together improve patient outcomes. Previous studies suggest that arsenic trioxide may enhance the efficacy of specific chemotherapy agents including those in DVd; however, research in people has not yet demonstrated this improved effectiveness. Because the safety of arsenic trioxide has been tested in this patient population, this phase II study will gather more information about safety and also measure efficacy through various measures.

Purpose: This study will evaluate the safety and efficacy of doxorubicin, vincristine and dexamethasone plus arsenic trioxide in untreated patients with symptomatic multiple myeloma. The biology of the tumor and other molecular changes will also be assessed in patients through collections of blood and marrow samples.

Treatment: Patients in this study will receive arsenic trioxide, doxorubicin, vincristine and dexamethasone. During the first five days of the study, patients will be given arsenic trioxide each day through an intravenous infusion. No treatments will be provided on days six and seven. After this first week, patients will then receive study drugs on the following schedule every four weeks: doxorubicin and vincristine on day one, dexamethasone on days one through four, and arsenic trioxide twice each week. This schedule can be repeated up to four times for a total of approximately four months. Several tests and exams will be given throughout the study to closely monitor patients. Supportive care will be provided to help regulate side effects from study drugs and maintain quality of life in patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have Multiple Myeloma
* No prior chemotherapy, thalidomide, or corticosteroids treatments for Multiple Myeloma
* ECOG performance status must be 0-2

Exclusion Criteria:

* Resting left ventricular cardiac ejection fraction ≥50% by echo or MUGA scan.
* QT interval ≥480 msec on baseline ECG.
* No history of cardiac disease.
* Pregnant or breast-feeding.
* No history of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the components of Doxil.
* History of prior or concurrent malignancy or myelodysplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07; Primary Completion 2006-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Assess the ability of DVd plus arsenic trioxide to achieve an overall response (complete and partial) rate in patients with untreated Multiple myeloma(MM) | 2004-2008

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Hofmeister CC, Jansak B, Denlinger N, Kraut EH, Benson DM, Farag SS. Phase II clinical trial of arsenic trioxide with liposomal doxorubicin, vincristine, and dexamethasone in newly diagnosed multiple myeloma. Leuk Res. 2008 Aug;32(8):1295-8. doi: 10.1016/j.leukres.2007.10.020. Epub 2007 Dec 21. PMID 18082257
- See also: Jamesline — http://cancer.osu.edu